CLINICAL TRIAL: NCT03821493
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE 2-PERIOD STUDY TO INVESTIGATE THE EFFECT OF MULTIPLE DOSES OF ITRACONAZOLE ON THE PHARMACOKINETICS OF A SINGLE DOSE OF PF-06651600 IN HEALTHY PARTICIPANTS
Brief Title: Effect of Multiple Doses of Itraconazole on the Pharmacokinetics of a Single-Dose of PF-06651600 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7981023; 2018-004664-55 (EudraCT Number)
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Healthy Participants
Keywords: PF-06651600; Itraconazole; CYP3A4; Drug-Drug Interaction
MeSH Terms: interventions — PF-06651600; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06651600 treatment arm (Experimental): This arm includes two treatment periods. Period 1-Single oral dose of PF-06651600 30 mg as tablets on Day 1 followed by Period 2 in which itraconazole 200 mg (oral solution) is given for 5 days. On Day 4 of Period 2, a single oral dose of PF-06651600 30 mg is given with itraconazole
  Interventions: Drug: PF-06651600 10 mg tablets; Drug: Itraconazole Solution 200 mg

INTERVENTIONS:
Drug: PF-06651600 10 mg tablets — On Day 1 in Period 1, a single oral dose of 30 mg (3 x 10 mg tablets) will be administered.
  On Day 4 of Period 2, a single oral dose of 30 mg (3 x 10 mg tablets) will be administered after itraconazole.
Drug: Itraconazole Solution 200 mg — Itraconazole 200 mg will be administered as 20 mL (10 mg/mL) oral solution once daily on Days 1-5 in Period 2.
  On Day 4 of Period 2, co-administration of itraconazole 200 mg and PF-06651600 30 mg will occur. Itraconazole will be administered first followed by PF-06651600 tablets.
  Other Names: Sporanox Oral Solution

SUMMARY:
This study will estimate the impact of a strong CYP3A4 inhibitor (itraconazole) on the pharmacokinetics of an investigational product (PF-06651600) in healthy adult participants.

This is an open-label, fixed sequence two period study with healthy participants that will receive a single dose of PF-06651600 alone and co-administered with multiple doses of itraconazole at a single center.

Participants will be screened within 28 days of the first dose of the investigational products and if entry criteria are met, the participant will report to the clinic on the day before the Day 1 visit. On Day 1 of Period 1, each participant will receive a 30 mg dose of PF-06651600 and PK samples will be collected for 48 hours. In Period 2, participants will receive itraconazole solution from Day 1-5. On Day 4 of Period 2 the participant will receive 30 mg of PF-06651600 with the itraconazole. PK samples will be collected up to 48 hours after the PF-06651600 dose. Participants will be confined for a total of 9 days in the clinic. The participant will be followed up by phone contact.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg.

Exclusion Criteria:

* Evidence of congestive heart failure or history of congestive heart failure or any of the following: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident including transient ischemic attack or pulmonary embolus.
* Known hypersensitivity to itraconazole or it excipients or to other azole antifungals.
* Infection with Hepatitis B, C or HIV
* Known present or history of malignancy other than a successfully treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Single dose Area under the curve from time zero to infinity [AUC (0-inf)] of PF-06651600 | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24 and 48 hours
  Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinity.
Maximum observed plasma concentration of PF-06651600 | 0, 0.5, 1, 2, 4, 6, 8, 12, 16, 24 and 48 hours
  Peak concentration of PF-06651600

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (AEs) | Baseline up to 35 days
Number of adverse events leading to discontinuation | Baseline up to 35 days
Number of participants with clinically significant change in vital signs from Baseline | Baseline to Day 9
Number of participants with clinically significant abnormalities in clinical laboratory values | Baseline to Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Be-bru, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981023&StudyName=A+PHASE+1%2C+OPEN-LABEL%2C+FIXED+SEQUENCE+2-PERIOD+STUDY+TO+INVESTIGATE+THE+EFFECT+OF+MULTIPLE+DOSES+OF+ITRACONAZOLE+ON+THE+PHARMACOKINETICS+OF+A+SINGLE+DOSE+OF+PF-06651600+IN+HEALTHY+PARTICIPANTS